CLINICAL TRIAL: NCT02994966
Title: Diabetes Foot Care Clinical Pathway - Orpyx Medical Technologies
Acronym: DFCCP-Orpyx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other); Orpyx Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AICE-201500873
Record Dates: First submitted 2016-12-09; First posted 2016-12-16 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surrosense (Experimental): Subjects randomized to this group will receive standard care, including appropriate off-loading and footwear as well as wear SurroSense Rx® in-shoe pressure-sensing arrays, which provide visual and auditory/vibratory feedback alerts (relating to high plantar pressures) and offloading guidance to a watch display intended to assist in the recurrence of diabetic foot ulcers. They will also be advised to perform daily self-checks of their feet for redness, callous and wounds. A daily checklist will be provided to participants to evaluate compliance.
  Interventions: Device: Surrosense
- Standard care (Active Comparator): Subjects randomized to this group will receive standard care, including appropriate off-loading and footwear. They will also be advised to perform daily self-checks of their feet for redness, callous and wounds. A daily checklist will be provided to participants to evaluate compliance.
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Surrosense
  Arms: Surrosense
Other: Standard care
  Arms: Standard care

SUMMARY:
In 2011, the premiers of all Canadian provinces and territories selected diabetes foot care as one of three significant targets for pan-provincial action. The Diabetes Foot Care Clinical Pathway Project (DFCCPP) aims to optimize methods of early detection and treatment of foot ulcers in an effort to reduce lower limb amputation (LLA) by 50%. The DFCCPP key deliverables apply consistency in assessment, care, treatment and process standards, early intervention and complex wound care management, while optimizing health outcomes. To achieve these deliverables, High Risk Foot Teams (HRFTs) will be implemented across the province starting with three pilot sites (Slave Lake, Brooks, and outpatient clinics at the Peter Lougheed Hospital). The pilot site facilities were selected on the basis of their employing staff with expertise and knowledge in diabetic foot care. The HRFT will assess and treat patients with moderate and high-risk findings, and this care pathway will then be rolled out to all clinicians who perform diabetic foot assessments (Primary Care, Home Care, Diabetes Centers, First Nations Reserves, etc.). In conjunction with the DFCCPP, we will evaluate the efficacy of a technological device developed by Alberta-based small-medium enterprise (SME) to improve diabetic foot outcomes by preventing future wounds in high-risk patients who have recently been treated for active foot ulcers. This technology is the SurroSense Rx® smart insole system (Orpyx Medical Technologies Inc., Calgary AB), a device that provides dynamic offloading guidance to patients, in addition to enabling ongoing adherence tracking by the HRFT. It is hypothesized that early wound detection and treatment will ultimately lead to improvements in wound prevalence, chronic wound care, and reduce the need for surgical intervention, including LLA.

DETAILED DESCRIPTION:
The Canadian Institute of Health Information estimates that foot wounds (with diabetes as the leading cause) are present in 4% of all hospital inpatients, 7% of homecare clients and 10% of long-term care (LTC) residents. Of 210,000 people with diabetes in Alberta, 5,250 will seek treatment of a foot ulcer annually. In Alberta in 2014-15 there were 425 LLAs performed on 309 diabetic patients representing an increase of 89 LLA over 2010-11. Moreover, there is a tremendous reduction in quality of life of the patients and attendant negative effects on their families. The 5-year mortality rate after a new-onset diabetic foot ulcer is 43-55%, and is as high as 74% for patients undergoing LLA.

Continuous monitoring of the diabetic foot and preventative foot care is of utmost importance for patients with diabetes. This is especially the case in high risk patients who have previously had foot ulcers. Improving and standardizing diabetic foot screening, early wound detection and treatment will ultimately lead to improvements in wound prevalence, chronic wound care, and the need for surgical intervention, including amputation.

Effective pressure offloading is a key tenet of diabetic ulcer prevention and care. The effectiveness of offloading interventions is intimately linked to the skin reperfusion that is seen when persistent external pressure is alleviated. Key modifiable parameters in mitigating tissue damage to the neuropathic foot are pressure and time. Exposures from 15 min to one hour at pressures greater than 240 mmHg, and from two hours or more at pressures greater than 67 mmHg, were found to cause cell death in rat muscle tissue. Despite this, there is limited information regarding the efficacy of interventions aimed at preventing pressure ulcers; a comprehensive review of the literature did not find enough evidence to recommend a repositioning frequency. A consensus document from an international review on pressure ulcer prevention states "patients confined to wheelchairs should be taught to reposition every 15 minutes".

While established pressure offloading interventions are able to statically reduce pressure on the active ulcer, they provide no dynamic relief of pressure. Since neuropathy is characterized by a loss of protective sensation (LOPS), the patient is often unaware of sustained pressure on a specific anatomic region over time. Even with static offloading instruments, it is conceivable that critical pressure and time thresholds can be dynamically exceeded without the patient's knowledge or ability to address the problem. Taken together, the literature provides support for a system that monitors pressure over time at key locations, and provides alert-based feedback to guide as-needed, patient-based offloading for use in patients with active ulceration.

Orpyx Medical Technologies Inc. (Orpyx), has developed a smart insole technology (the "SurroSense Rx®") that senses pressure points in the user'splantar foot. This is important because pressure "hot spots" can lead to wound development that, if left untreated, can progress to a foot ulcer and LLA. Individuals able to maintain lower in-shoe peak pressures had 60% lower risk of foot ulcer recurrence. Unpublished studies with this device are demonstrating an 83% relative risk reduction in plantar ulceration in active versus control arms. This device provides dynamic offloading guidance to patients, in addition to enabling ongoing adherence tracking. This device has been shown to be an effective treatment in the management of diabetic foot patients at risk for ulcers, with respect to the care of active ulcers, in addition to prevention of future recurrence. Wearers of the SurroSense Rx® technology are provided with on demand cues for offloading, and should therefore have enhanced responsiveness and self-control over their foot care, thereby leading to a reduction in re-ulcerative events and thus, LLA.

The SurroSense Rx® system is a patent pending (US Publication 20120109013 and PCT WO/2012/055029) footwear system intended to prevent first and recurrent plantar ulcers, and to treat active ulcers in neuropathic patients. It comprises two pressure-sensing inserts and a smartwatch display device. The device alerts the user when "safe" pressure and time thresholds have been exceeded; the current thresholds are based on the results of a comprehensive review of the literature, which indicates that a conservative threshold would be >30-50mmHg for >15 minutes. As more plantar pressure and outcome data are collected over time, these thresholds may be modified as need be. The device measures plantar pressures at discrete points corresponding to bony prominences that would be considered to be at higher risk for ulceration: the first metatarsal head (1), the lateral metatarsal heads (2), the great toe (1), the lateral toes (1), the lateral foot (2), and the heel (1). These areas were selected based on the inherent high risk of neuropathic ulceration at these anatomic locations. This data is tracked, with analysis being performed on those that have been collected over the last 15 minutes. If > 95% of the measurements taken by a pressure sensor over a 15-minute scanning window exceed 30-50 mmHg, an alert is sent to the user via the smartwatch to guide them to appropriately offload that area.

The SurroSense Rx® device will be used as an adjunct in the treatment pathway following closure of diabetic foot wounds. It is widely acknowledged that, following wound healing, 50-100% of diabetic foot ulcers recur over a five-year period. What is more, it is estimated that after 18 months, 42% of ulcers recur, with half of those recurring in the first six months. Thus, it is the first six months following wound healing that is the most sensitive time for recurrence of ulceration. It is this critical patient population that will be fitted with the SurroSense Rx® device for secondary prevention of ulceration.

Taken together, diabetes patients with foot wounds are at an elevated risk of infection and LLA. Therefore, there is a need for an effective tool for the prevention and management of the diabetic foot.

Research Question and Objectives:

Does improving and standardizing foot screening for diabetes patients through the DFCCP concurrently with the use of the SurroSense Rx® smart insole system reduce the proportion of foot ulcer recurrence compared to patients who are receiving standard care? The objective of this proposal is to demonstrate that when combined with the DFCCP, the SurroSense Rx® smart insole system device is an effective modality that is superior to the current standard of care for preventing the recurrence of healed pressure ulcerations on the feet of subjects with diabetic peripheral neuropathy of the lower extremities. It is hypothesized that the use of the device will lead to a reduction in the risk of pressure ulcer recurrence in the Intervention group and to improve those subjects' foot self-care, when compared to subjects in the Control group. Over the longer term we anticipate that use of the technology in concert with the DFCCP will result in better foot health for diabetic patients. The ability to test the efficacy of the SurroSense Rx® device in parallel with the DFCCP implementation will allow the evaluation in a real-world setting where patients also have access to HRFT for prescription of the device. High Risk Foot Teams will be implemented across the province starting with three pilot sites (Slave Lake, Brooks, and the Diabetic Foot and Limb Preservation Centre at the Peter Lougheed Hospital), These pilot sites will be selected as facilities have existing staff with expertise and knowledge in diabetic foot care. The HRFT will assess and treat patients with moderate and high-risk findings. The AICE-funded project is a sub-study. All patients are clinically assessed in a standardized manner using the Alberta Foot Risk Assessment Form (AFRAF), which incorporates a standardized wound assessment and treatment approach.ces, ongoing assessment and embedded evaluation.

ELIGIBILITY:
Inclusion Criteria:

* History of diabetic foot ulcer that has resolved within the past twelve (12) months

  * Sensory abnormality with no skin breakdown/ulcer
  * Diabetes (according to AAFP diagnostic criteria (8))
  * Absent sensation to 10 g monofilament exam at 1 or more sites
  * Age >18y
  * One or more pedal pulses palpable or doppler-able on each foot (dorsalis pedis & posttibialis)
  * Ability to understand the use of the technology
  * Life expectancy greater than the duration of the study
  * Subject is willing and able to maintain the required offloading (as applicable for the location of the ulcer)
  * Subject or responsible caregiver is willing to adhere to the routine calibration schedule required for the proper ongoing functioning of the device (i.e., going through a monthly two minute procedure)
  * Has footwear that is compatible with the Orpyx device: diabetic shoes, running shoes, walking shoes; either lace-up or Velcro; must have a removable insert or orthotic

Exclusion Criteria:

* Weight > 325 lb (147 kg)
* Uncorrected visual impairment
* Active plantar ulceration or skin breakdown
* Presence of severe schema (absence of palpable or dopplerable foot pulses)
* Active Infection
* Abnormal toe, ankle and/or foot range of motion that would preclude the patient's ability to offload pressure alerts
* Gross foot deformity that would impact anatomical plantar pressure distribution (i.e., including Charcot foot deformity, and/or previous partial or complete foot or ray amputation)
* Insoles or orthotics with a hard plastic, or uneven, undersurface
* Patient is being cared for exclusively via Telehealth (i.e. there is no opportunity for hands-on or face-to-face interaction between the patient and the caregiving team)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Foot ulcer recurrence | 12 months
  hazard ratio

SECONDARY OUTCOMES:
Time to re-ulceration | 12 months maximum
Patient satisfaction | Last visit to High Risk Foot Team (maximum 12 months)
  Survey
Patient compliance | Last visit to High Risk Foot Team (maximum 12 months)
  Survey
Clinical adoption | 12 months
  Interviews with clinicians
Cost effectiveness | 12 months
Complications rates | 12 months
  new ulceration, ulcer extension, infection, surgical intervention, amputation, hospitalization documented
Determinants of ulcer formation | 12 months
  Pressure and adherence parameters compared with area of ulceration

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Brooks Home Care, Brooks, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - Slave Lake Family Care Clinic, Slave Lake, Alberta

IPD SHARING:
Plan to Share IPD: No